CLINICAL TRIAL: NCT02080390
Title: Strain Imaging in Breast Cancer Patients Receiving Trastuzumab
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201300763
Record Dates: First submitted 2014-02-27; First posted 2014-03-06 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Her 2 Positive Breast Cancer
Keywords: Her 2 Positive Breast Cancer; Trastuzumab; Herceptin; Heart Failure; Echocardiography
MeSH Terms: conditions — Heart Failure | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transthoracic echocardiogram (ultrasound): Any transthoracic echocardiogram (ultrasound) of the heart, performed as part of standard clinical care, will be further evaluated for special parameters that may help to detect weakening.
  Interventions: Procedure: Transthoracic echocardiogram (ultrasound)

INTERVENTIONS:
Procedure: Transthoracic echocardiogram (ultrasound) — Any transthoracic echocardiogram (ultrasound) of the heart, performed as part of standard clinical care, will be further evaluated for special parameters that may help to detect weakening.
  Other Names: Transthoracic echocardiogram

SUMMARY:
The purpose of this research study is to evaluate the effects of the chemotherapeutic drug, Trastuzumab (Herceptin) on the heart. Trastuzumab (Herceptin) is used to treat specific types of breast cancer and is known to cause weakening of the heart. Unfortunately, little is know as to why this this happens. The investigators want to identify any factors that may lead to the early detection, treatment and prevention of the cardiotoxicity (heart problem) associated with this drug.

DETAILED DESCRIPTION:
As a subject participating in this study the following information will be collected: complete past medical history including age, height, and weight will be done with each echocardiogram; blood pressure at clinic visits during treatment with trastuzumab, type of cancer will be noted, type of chemotherapy, doses of chemotherapy, type and dose of chemotherapy in the past, type and dose of radiation therapy received, names and doses of cardiac medications, results of cardiac tests, results of lab tests, family history of heart disease, and social history which will include risk factors for developing heart disease including tobacco and alcohol use. This information will be entered into a database for the investigators to try and detect any factors that may lead to the cardiotoxicity (heart problem) that may be caused by Trastuzumab (Herceptin).

Any transthoracic echocardiogram (heart ultrasound) ordered will be further evaluated for special parameters that may help to detect weakening of the heart earlier than a normal ultrasound. An echocardiogram (heart ultrasound) is when a probe is placed on the chest and pictures are taken using sound waves and a special camera.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Her 2 positive breast cancer.
* Patients who are currently receiving Trastuzumab (Herceptin).
* Patients who received Trastuzumab (Herceptin) after the formation of the UFHealth Medical Plaza pharmacy database was initiated.

Exclusion Criteria:

* Age less than 18 years
* Patients who have not received Trastuzumab (Herceptin).
* Patients who received Trastuzumab prior to the formation of the UFHealth Medical Plaza pharmacy database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women or men recieveing Trastuzumab (Herceptin) for HER2 positive breast cancer.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10-28 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Longitudinal Strain | Change in baseline longitudinal strain from beginning of study to end of study. Patients will be followed for a minimum of 1 year.
  Each transthoracic echocardiogram obtained during the patient's treatment will be assessed for longitudinal strain.
Left Ventricular Ejection Fraction | Change in ejection fraction from baseline to end of study. Patients will be followed for a minimum of 1 year.
  Left ventricular ejection fraction from all clinically indicated transthoracic echocardiograms will be compared from baseline through the end of the study.

SECONDARY OUTCOMES:
Clinically evident congestive heart failure | From baseline to end of study. Patients will be followed for a minimum of 1 year.
  Clinically evident congestive heart failure(symptoms of fluid overload such as shortness of breath, dyspnea on exertion, orthopnea or paroxysmal nocturnal dyspnea or physical findings of congestive heart failure such as jugular venous distension, rales on pulmonary exam, lower extremity edema).
Cardiac medication use | Baseline to end of study. Patients will be follwed for a minimum of 1 year.
  The type and dose of all cardiac medications will be followed from baseline to end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hamburger, DO, MPH, Principal Investigator — University of Florida
Locations (1):
- Univerisity of Florida, Gainesville, Florida, United States